CLINICAL TRIAL: NCT07034001
Title: Effect of Anesthesia on Frontal QRS-T Angle in Obese Individuals
Brief Title: Effect of Anesthesia on Frontal QRS t Angle in Obese Individuals
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Harun Tolga Duran, Ass. Prof., Amasya University
Other Study IDs: htdekg
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity; frontal qrs-t angle
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BMI>30: BMI>30
- BMI<30: BMI<30

SUMMARY:
The aim of this observational study is to determine the effect of anesthesia on frontal qrs-t angle changes in obese individuals. To learn the long-term effects of intervention A in individuals with a body mass index > 30 who received intervention A. The main question it aims to answer is:

Does frontal qrs-t angle change occur in obese individuals due to anesthesia? Preoperative and intraoperative ECG changes of individuals undergoing surgery will be examined.

DETAILED DESCRIPTION:
All patients were routinely administered 500 cc of Ringer's lactated solution intravenously (IV) before anesthesia and taken to the operating room. The body mass index will be calculated according to the formula body weight kg / height cm2. Obese patients with a BMI above 30 kg/m2 were recorded as group 2, and non-obese patients with a BMI below <30 kg/m2 were recorded as group 1. Patients were taken to the operating room and routine ECG, noninvasive blood pressure, pulse, and oxygen saturation monitoring (CARESCAPE™ B650, GE Healthcare, USA) was performed. All patients were hydrated intravenously (IV) with 500 cc of Ringer's lactated solution after a 6-hour fast. For premedication, midazolam 1 mg IV and pantoprazole 40 mg IV were administered. For anesthesia induction, propofol 2 mg/kg, fentanyl 2 mg/kg and rocuronium 0.6 mg/kg were administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 18-65 who underwent laparoscopic cholecystectomy surgery

Exclusion Criteria:

* known coronary artery disease, atrial fibrillation, heart failure, liver failure, kidney failure, preexcitation syndromes, electrolyte disorders, use of drugs that prolong the QT interval, respiratory failure and metabolic diseases were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People between the ages of 18-65 who underwent laparoscopic cholecystectomy surgery
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
EKG | 1 day
  Frontal qrs t angle and qt interval examination on ecg
Frontal qrs-t angle | 1 day
  Frontal qrs t angle examination on ecg

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
single-center study

REFERENCES:
- [Result] Kaya A, Karahan MA, Bingol Tanriverdi T, Esercan A, Bostanci Erkmen M, Tanriverdi Z. Comparison of the Effects of Spinal Anaesthesia on Frontal QRS-T Angle in Term and Post-Term Pregnancies Planned for Elective Caesarean Section: A Prospective Study. Medicina (Kaunas). 2025 May 19;61(5):919. doi: 10.3390/medicina61050919. PMID 40428877